CLINICAL TRIAL: NCT05351021
Title: Efficacy of Metformin as Preventive Treatment in Paclitaxel Induced Peripheral Neuropathy in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Principal investigator-Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-375
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Neuropathy; Breast Cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (metformin group) (Experimental): who will receive adjuvant paclitaxel in addition to metformin tablets (1700 mg daily) during the chemotherapy treatment duration.
  Interventions: Drug: Metformin
- Group II (control group) (Placebo Comparator): who will receive adjuvant weekly paclitaxel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — cidophage 850 gm twice daily
  Arms: Group I (metformin group)
Drug: Placebo — placebo twice daily for treatment period
  Arms: Group II (control group)

SUMMARY:
At present, there are no FDA-approved treatments for chemotherapy-induced neuropathy. Discrete neuro anti-inflammatory effects of metformin support its repurposing as a neuroprotective agent in patients with neurodegenerative diseases. Therefore, this study aims to evaluate the effect of metformin on the amelioration of paclitaxel induced neuropathy in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Early-stage breast cancer patients who will receive adjuvant paclitaxel
* Performance status according to Eastern Cooperative oncology group (ECOG) < 2.
* Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count ≥100,000/mm3), liver function (serum total bilirubin <1.5 mg/dl), renal function (creatinine<1.5 mg/dl).

Exclusion Criteria:

* Clinical neuropathy at prior to enrollment.
* Patients treated with medications that increase the risk of neuropathy like amiodarone, Colchicine, metronidazole, phenytoin.
* Patients with a history of hypersensitivity to metformin.
* Pregnant or lactating females.
* Patients who are using metformin for any other cause.
* Patients with Diabetes mellitus.
* Receiving vitamin B1, B6, B12 or another vitamin supplemental therapy.
* Receiving antidepressants, opioids, adjuvant analgesic agents (eg, anticonvulsants, clonazepam, or mexiletine), topical analgesics, and amifostine.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The incidence of grade II or more peripheral neuropathy at the end of paclitaxel treatment | 8 weeks
  Grading of paclitaxel induced peripheral neuropathy will be done using NCI-CTCAE version (4.03)

SECONDARY OUTCOMES:
Time to develop grade 2or 3 PIPN | 8 weeks
  The time from randomization till development of grade II or III PN will be recorded for all patients included in the study.
the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity(FACT-GOG-NTX) subscale | 8 weeks
  Patient's QOL will be assessed using the validated Arabic version of FACT-GOG-NTX subscale
Pain Severity | 8 weeks
  The severity of neuropathic pain will be assessed using the Arabic version of the Brief Pain Inventory Short Form (BPI-SF)
Serum biomarkers level in (ng/mL) | 8 weeks
  Nerve growth factor Biomarkers levels will be measured using commercial ELISA kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Bakry HM, Mansour NO, ElKhodary TR, Soliman MM. Efficacy of metformin in prevention of paclitaxel-induced peripheral neuropathy in breast cancer patients: a randomized controlled trial. Front Pharmacol. 2023 Jul 31;14:1181312. doi: 10.3389/fphar.2023.1181312. eCollection 2023. PMID 37583905